CLINICAL TRIAL: NCT07095556
Title: Impact of Nd: YAG Laser Photobiostimulation on Healing of Gingiva Following Tooth Extraction and Alveolar Ridge Preservation
Brief Title: Impact of Nd:YAG Laser Photobiostimulation on Healing of Gingiva
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00139090
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Wound Healing and Prevention; Oral Inflammation; Photobiomodulation; Post-operative Pain Management; Tooth Extraction Site Healing
Keywords: Inflammation; Periodontal Disease; low-level laser therapy; gingival healing; Post-operative pain
MeSH Terms: conditions — Inflammation; Periodontal Diseases; Pain, Postoperative | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Sham laser will be applied instead of the low-level laser.
- Intervention (Experimental): Low-level lase therapy will be applied at tooth extraction sites.
  Interventions: Other: Low-level laser therapy

INTERVENTIONS:
Other: Low-level laser therapy — The low-level laser applications will be made on the same day as the standard of care treatment (day 1), and then day 3, and day 7 by a study team member who is trained in the use of the laser device.
  The laser photobiostimulation will be applied using LightWalker® laser (FOTONA), with following settings, Nd:YAG laser 1064 nm, MSP modality (pulse duration), 0.5 W (power), 10 Hz (frequency), 1 min/ 1 cm2 spot using Genova handpiece from buccal, lingual, and occlusal aspects. The Genova handpiece will be placed 1 cm away from gingival tissue.
  Participants and operators will wear glasses to protect their eyes from laser beam in all sessions.
  Arms: Intervention

SUMMARY:
The intervention in this study is to determine whether multiple applications of photobiostimulation with Nd-YAG laser improve wound healing following tooth extraction and alveolar ridge preservation. Investigators plan to assess the impact of laser treatment on wound healing by measuring salivary biomarkers, gingival wound size and surveying for the use of pain reduction and patient satisfaction. The intervention group will receive extraction and alveolar ridge preservation with Nd-YAG laser photobiostimulation on days 1, 3, and 7 following extraction and socket preservation, while the control group will receive the standard of care extraction and alveolar ridge preservation without the laser

DETAILED DESCRIPTION:
Photobiostimulation, also known as low-level laser therapy (LLLT) or phototherapy, utilizes a low-level laser to increase cell proliferation, enhance cell stimulation, and reduce gingival inflammation. It has been reported that photobiostimulation enhances chemical and metabolic changes and alters cellular behavior in the tissue by light absorption. Photobiostimulation as an adjunct treatment modality can accelerate the healing process, improve patient comfort and satisfaction following dental surgical procedures, and benefit patients with compromised healing capacity.

Alveolar ridge preservation (ARP) is a standard procedure to minimize alveolar bone and gingival soft tissue atrophy following tooth extraction and before dental implant placement. The healing of ARP is critical for the success of implant placement timely treatment. The ARP procedure is currently the standard practice for patients interested in dental implant treatment and involves bone grafting of the extracted socket. ARP techniques have been used for over 20 years to maintain a favorable soft and hard tissue morphology for dental implant-related restorations.

The purpose of this study is to understand the impact of Nd-YAG laser photobiostimulation on wound healing when combined with tooth extraction and alveolar ridge preservation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are ≥ 18 years old,
* Patients who are scheduled for the treatment of tooth extraction and alveolar ridge preservation (ARP)
* No contraindications for tooth extraction and alveolar ridge preservation based on electronic health records.
* Participants who can express the level of pain
* Participants who self-report "not pregnant"

Exclusion Criteria:

* Untreated periodontal disease
* Acute infection of the teeth
* Use of antibiotics within the last three months.
* Pregnant or lactating women
* Use of bisphosphonates based on EHR
* Alveolar bone defects occurred or were detected during tooth extraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers in saliva | From day of tooth extraction through day 7
  The measurement of inflammatory and anti-inflammatory markers in saliva, IL-1β, IL-6, IL-8, IL-10, IL-12 and TNF secreted during the early stages of wound healing at day 3 and day 7.
Wound size dimensional changes | From the day of tooth extraction to day 42
  The comparison of dimensional changes in wound size between test and intervention groups. Digital gingival scans of the wound will be taken immediately after surgery and at days 3, 7, 14, and 42 for Aim 2.
Post-operative pain | From post-operative day 3 to day 14
  Recording of pain perception using a Visual Analog Scale at visits 3, 7, and 14 (maximum pain being 10 vs. no pain being 0), 2)

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Emecen-Huja, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC College of Dental Medicine, Graduate Periodontics Clinic, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keskiner I, Lutfioglu M, Aydogdu A, Saygun NI, Serdar MA. Effect of Photobiomodulation on Transforming Growth Factor-beta1, Platelet-Derived Growth Factor-BB, and Interleukin-8 Release in Palatal Wounds After Free Gingival Graft Harvesting: A Randomized Clinical Study. Photomed Laser Surg. 2016 Jun;34(6):263-71. doi: 10.1089/pho.2016.4094. Epub 2016 Apr 18. PMID 27088277
- [Background] Cafiero C, Spagnuolo G, Marenzi G, Martuscelli R, Colamaio M, Leuci S. Predictive Periodontitis: The Most Promising Salivary Biomarkers for Early Diagnosis of Periodontitis. J Clin Med. 2021 Apr 3;10(7):1488. doi: 10.3390/jcm10071488. PMID 33916672
- [Background] Saglam M, Koseoglu S, Tasdemir I, Erbak Yilmaz H, Savran L, Sutcu R. Combined application of Er:YAG and Nd:YAG lasers in treatment of chronic periodontitis. A split-mouth, single-blind, randomized controlled trial. J Periodontal Res. 2017 Oct;52(5):853-862. doi: 10.1111/jre.12454. Epub 2017 Mar 23. PMID 28332191
- [Background] Fulop AM, Dhimmer S, Deluca JR, Johanson DD, Lenz RV, Patel KB, Douris PC, Enwemeka CS. A meta-analysis of the efficacy of laser phototherapy on pain relief. Clin J Pain. 2010 Oct;26(8):729-36. doi: 10.1097/AJP.0b013e3181f09713. PMID 20842007
- [Background] Mizutani K, Aoki A, Coluzzi D, Yukna R, Wang CY, Pavlic V, Izumi Y. Lasers in minimally invasive periodontal and peri-implant therapy. Periodontol 2000. 2016 Jun;71(1):185-212. doi: 10.1111/prd.12123. PMID 27045437
- [Background] Krizaj Dumic A, Pajk F, Olivi G. The effect of post-extraction socket preservation laser treatment on bone density 4 months after extraction: Randomized controlled trial. Clin Implant Dent Relat Res. 2021 Jun;23(3):309-316. doi: 10.1111/cid.12991. Epub 2021 Mar 8. PMID 33686771